CLINICAL TRIAL: NCT05145647
Title: To Observe the Local Tumor Recurrence Rate of Adding Intraluminal Brachytherapy With Balloon Applicator After Standard Definitive Concurrent Chemoradiotherapy (CCRT) on Local-regional Thoracic Esophageal Cancer Patients Who Refused Surgery
Brief Title: To Observe the Benefit of Adding Brachytherapy After CCRT on Resectable Esophageal Cancer Patients Without Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202100288A3
Record Dates: First submitted 2021-09-03; First posted 2021-12-06 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-07

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Add-on Brachytherapy (Experimental): The evaluation for feasibility of surgery takes place 5-6 weeks after CCRT. Any subject whose tumor status is resectable at evaluation but declines surgical proposal will be eligible to be enrolled in the following study phase.
  Interventions: Radiation: Add-on Brachytherapy; Device: "BRAXX" Esophageal Brachytherapy Applicator

INTERVENTIONS:
Radiation: Add-on Brachytherapy — Brachytherapy protocol starts within 2 weeks after consolidative EBRT, subjects who are enrolled will receive brachytherapy with specified balloon applicator. High-dose-rate (HDR) brachytherapy system will be used in the treatment, 5-Gy per fraction is delivered to the pre-treatment esophageal length of primary tumor(s), second treatment if applicable will be finished within 2 weeks after the first one, a total of 5-10Gy in 1-2 fractions will be delivered.
Device: "BRAXX" Esophageal Brachytherapy Applicator — The device is intended for use with commercially available afterloader during brachytherapy. The purpose of the device is for delivery of radioactive source to the esophagus. This device is sterile, disposable and single-use.
  Other Names: 510(K) Number: K183332 (class II)

SUMMARY:
Clinical experience of adding intraluminal brachytherapy with traditional applicator after definitive concurrent chemoradiotherapy (CCRT) for local-regional thoracic esophageal cancer is limited due to high complication risk and non-superiority in survival. The innovative applicator can maximize the therapeutic efficacy by reducing dose inhomogeneity in the esophageal wall, which will translate into less over-dosing and less risk of the side effects of fistula or stenosis.

The primary goal of this study by using new applicator is to observe the change in local tumor control rate, while secondary goals are treatment related toxicity, progression-free survival, and overall survival.

DETAILED DESCRIPTION:
American Brachytherapy Society (ABS) provided guidelines for brachytherapy in esophageal cancer in 1997, which defines the general principle for brachytherapy used in definitive CCRT. (1) Patients with unifocal thoracic adeno- or squamous cancers < or = 10 cm in length, with no evidence of intra-abdominal or metastatic disease.

(2) Contraindications include tracheal or bronchial involvement, cervical esophagus location, or stenosis that cannot be bypassed.

(3) The esophageal brachytherapy applicator should have an external diameter of 6-10 mm.

(4) If 5FU-based chemotherapy and 45-50-Gy EBRT are used, recommended brachytherapy is HDR 5-10 Gy in one to two weekly fractions of 5 Gy each and should not be given concurrently with chemotherapy In the esophageal cancer treatments, tumor recurrence in the primary tumor site approaches 50% in most non-surgical CCRT series reported. Brachytherapy has the advantages of introducing higher doses to the tumor site to improve tumor control, but it is like the double edge of the sword, higher dose may bring higher risk of serious side effect, such as fistula formation in the esophagus noted over previous studies. The innovative Braxx applicator can maximize the therapeutic efficacy by reducing dose inhomogeneity in the esophageal wall (3mm to surface: 136-175%), which will translate into less over-dosing and less risk of the side effects of fistula or stenosis as noted in traditional brachytherapy using NG tube (3mm to surface: 160%-265%). Without much changing the user's habits in performing brachytherapy, the innovative applicator is expected to be easier to be accepted for use.

* Screening Phase: All non-T4b or M1 (non-nodal organ involvement) stage esophageal cancer participants who received neoadjuvant/ definitive chemoradiation first, which includes radiotherapy dosage between 4140-5040cGy concurrently with chemotherapy of carboplatin + paclitaxel or cisplatin + 5FU.

* The evaluation for feasibility of surgery takes place 5-6 weeks after CCRT. Any participant's tumor status is resectable at evaluation but declines surgical proposal will be eligible to be enrolled in the following study phase.
* Eligible participant receives consolidative CCRT, which includes EBRT dosage of 2000cGy concurrently with chemotherapy of carboplatin + paclitaxel or cisplatin + 5FU as the investigators' status quo.

  * Brachytherapy Study Phase:

Brachytherapy protocol starts within 2 weeks after consolidative EBRT (This is "Week 1"), enrolled participants will receive brachytherapy with specified balloon applicator. High-dose-rate (HDR) Nucletron brachytherapy system will be used in the treatment, 5-Gy per fraction is delivered to the pre-treatment esophageal length of primary tumor(s), second treatment if applicable will be finished within 2 weeks after the first one, a total of 5-10Gy in 1-2 fractions will be delivered.

The distance from the center of radiation source to the surface of applicator is 6-9mm depending on the air volume inflated into the balloons in the applicator, the esophageal mucosa will be attached against to the surface of inflated balloon, radiation dose prescribed at 3mm away from the balloon surface will cover most of the esophageal wall, and 5Gy will be prescribed there. Efforts will be made to reduce the high dosage volume in adjacent normal organs, also to reduce the hot spot within treated esophageal wall. It is NOT allowed to give concurrent chemotherapy on the days of HDR brachytherapy. Grade 3 and higher grade toxicity may cause a prolonged interval between the two brachytherapy treatments, either dose reduction or delay treatment according to tolerability of individual participant is allowed. If participant can't tolerate full course of brachytherapy, the total dose (EBRT+brachytherapy) can be reduced to 25Gy without violation of protocol. The management of adverse effects will follow general principles.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 20-85 years, with ECOG performance 0-2
2. Thoracic esophageal cancer with clinical stage I-III and biopsy proof; patient with cervical esophageal cancer or stage IV thoracic esophageal cancer could be recruited in this trial according to Investigator's assessment.
3. Complete first course CCRT with minimum doses of 40 Gy to tumor and nodal area via external beam radiotherapy (EBRT).
4. Patient whose tumor is resectable but declined to receive surgery after first course CCRT.

Exclusion Criteria:

1. T4b tumor status (tracheal / bronchial mucosa, aortic involvement, or fistula formation).
2. Stenosis of esophageal lumen that cannot be bypassed by the applicator.
3. The primary tumor length exceeds 20cm.
4. The patient is participating in other clinical trials.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2025-06-18 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
To estimate the local control rate at primary tumor site | 12 months after completion of treatment
  Enrolled subject will be followed every 3 months after treatment, EGD-endoscope (± biopsy) will be arranged at Month 3, 6, 9, 12 and CT scans on Month 6, 12, to evaluate the tumor status.

SECONDARY OUTCOMES:
Treatment toxicity grading according to the CTCAE | 12 months after completion of treatment
  Treatment toxicity will be recorded at each visit as CTCAE v5.0.

OTHER OUTCOMES:
Progression-free survival (PFS) | 12 months after completion of treatment
  the tumor status or patient's survival status within 1 year after treatment
Overall survival (OS) | 12 months after completion of treatment
  patient's survival status within 1 year after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chen-Kan Tseng, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Linkou Chang Gung Memorial Hospital, Taoyuan, Taiwan